CLINICAL TRIAL: NCT05057585
Title: The Effects of Bed Exercises on Anxiety, Pain, Early Ambulation and Mobilization in Patients
Brief Title: The Effects of Bed Exercises on Anxiety, Pain, Early Ambulation and Mobilization in Patients Undergoing Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gurkan Kapikiran (Other)
Responsible Party: Sponsor-Investigator, Gurkan Kapikiran, Assistant Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2020/33
Record Dates: First submitted 2021-09-03; First posted 2021-09-27 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Surgery; Anxiety; Pain
Keywords: Anxiety; Early ambulation; Bed exercise; Major surgery; Mobilization
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Beds

STUDY DESIGN:
Intervention Model Description: This research was conducted as a prospective and experimental study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Each patient in the experimental group was given in-bed exercises for 15 minutes. An anxiety questionnaire was asked to both the experimental and control groups. It was expected that both the experimental and control group patients would be stable in the postoperative period. The same exercises were applied again for 15 minutes to the patients who were stable after the surgery. Then the patients were made to take steps around the bed. Pain levels were measured.
  Interventions: Behavioral: Turning in bed, arm and leg exercises
- No treatment group (No Intervention): Apart from clinical protocols, no application was made in patient follow-up. Anxiety scale was filled and pain level was evaluated. Pain and anxiety scales were refilled within the same period without any application.

INTERVENTIONS:
Behavioral: Turning in bed, arm and leg exercises — Exercises (arm and leg exercises, turning in bed) were applied only to the experimental group. It was applied for 15 minutes 12-24 hours before the operation.
  Arms: Exercise group

SUMMARY:
In this study, the effects of bed exercises on pain, anxiety, early ambulation and mobilization in major surgery patients were aimed. The research was experimental and a total of 120 patients participated. Data were collected using an information form, anxiety scale, and pain scale. Exercise was applied to the patients in the experimental group (15 minutes) and no intervention was applied to the control group. Descriptive statistics, correlation tests and t-test were used. Cronbach's alpha coefficients were checked for the scales.

DETAILED DESCRIPTION:
Major surgery are operations that can cause morbidity and mortality. Worldwide, approximately 230 million major surgical interventions are performed each year. Major surgery is a stressful experience and causes life-threatening fear and anxiety by increasing the level of anxiety. The most important of these fears is the pain that may occur after surgery. More than 75% of patients who experience postoperative pain in the Western world report that they experience moderate to severe pain. In our country, this rate is over 90%. If pain management is inadequate, patients' quality of life is adversely affected. In pain management, nurses can use non-pharmacological methods such as massage and exercise in addition to pharmacological applications.

Leg-arm exercises done in bed are aimed at protecting the muscle strength of individuals. Turning in bed, leg-arm exercises, raising the heels and feet, inverting the arms, moving from right to left, reverse arm and leg movements are performed. Also 6-8. Early ambulation is recommended. If these applications are made, early recovery and rapid discharge can be achieved. Since pain and anxiety delay early recovery in patients undergoing major surgery, effective pain management is very important. In this study, we aimed to examine the effects of in-bed exercises on anxiety and pain in patients undergoing major surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Ability to communicate verbally and not having a cognitive problem,
* Defining pain severity of 4 and above,
* Willing to participate in the study,
* Having undergone major surgery.

Exclusion Criteria:

* The absence of open wounds and cellulite in the area to be applied,
* The absence of thrombophlebitis,
* The absence of deep vein thrombosis,
* The absence of inflammatory diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Anxiety | 0-15 minutes
  It is the form in which the patient's anxiety is measured. The expected value in the scale is between 0 and 50 points. As the Scale Score increases, the level of anxiety also increases.
Pain level | 0-15 minutes
  It is a measure of pain level. Pain intensity ranges from 0 to 10, 0 points no pain, 10 points unbearable pain.
Early Ambulation | 0-15 minutes
  It is the form in which the postoperative mobilization times are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No